CLINICAL TRIAL: NCT02197585
Title: Cyanoacrylate vs Suture for Mesh Fixation in Inguinal Hernia Surgery
Brief Title: Comparison of Mesh Fixation Wit Cyanoacrylate vs Suture in Inguinal Hernia Surgery
Acronym: UHU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital del Mar (Other)
Responsible Party: Principal Investigator, José A. Pereira, Medico Adjunto Cirugia General, Hospital del Mar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UHU
Record Dates: First submitted 2014-07-21; First posted 2014-07-22 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Pain
Keywords: Male patients; Age > 18 year; Primary hernia; glue
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glue (Experimental): Mesh fixation with glue
  Interventions: Procedure: Inguinal mesh hernioplasty
- Suture (Active Comparator): Mesh fixation with suture
  Interventions: Procedure: Inguinal mesh hernioplasty

INTERVENTIONS:
Procedure: Inguinal mesh hernioplasty

SUMMARY:
To compare fixation with glubran2 with suture during surgery por primary inguinal hernia.

Hypothesis: Glue may induce less complications and chronic pain than suture

ELIGIBILITY:
Inclusion Criteria:

* Male patients
* Aged more than 18 years
* Primary inguinal hernia

Exclusion Criteria:

* Inguinoscrotal hernia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2007-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Chronic pain after two years | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: JA Pereira, MD, Principal Investigator — Hospital del Mar